CLINICAL TRIAL: NCT04843670
Title: Modified Pancreaticojejunostomy Technique With Isolated Pancreatic Loop After Pancreaticoduodenectomy Reduces Postoperative Pancreatic Fistula: a Retrospective Study
Brief Title: Isolated Pancreatic Loop With Modified Pancreaticojejunostomy
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, clinical professor, Université de Sousse
Other Study IDs: U23471
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Pancreaticoduodenectomy
Keywords: Pancreaticoduodenectomy; pancreaticojejunostomy; Postoperative pancreatic fistula.
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients operated for pancreas tumors: duodenopancreatectomy for head of the pancreas tumors
  Interventions: Procedure: duodenopancreatectomy

INTERVENTIONS:
Procedure: duodenopancreatectomy — resection of the head of the pancreas, the mower part of the biliary duct, and antrectomy

SUMMARY:
The aim of the present study was to observe whether the modified pancreatico- jejunostomy (PJ ) technique with an isolated pancreatic loop would effectively reduce the POPF rate and overall morbidity after PD

DETAILED DESCRIPTION:
Postoperative pancreatic fistula (POPF) is widely regarded as the most threatening complication following pancreaticoduodenectomy (PD). Its clinical impact and sequelae have been previously described and shown to contribute to the development of other morbid complications and high rates of mortality.

The aim of the present study was to observe whether the modified pancreatico- jejunostomy (PJ ) technique with an isolated pancreatic loop would effectively reduce the POPF rate and overall morbidity after PD.

Methods: We report our early experience using a modified PJ technique with an isolated pancreatic loop after after PD in 201 patients between January 2010 and December 2020.

ELIGIBILITY:
Inclusion Criteria:

* age up to 30
* head of the pancreas tumor

Exclusion Criteria:

* body and tail pancreatic tumors

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing duodenopancreatectomy procedure, in the surgery department .
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of pancreatic fistula | 10 years
  level of lipase in abdominal drain after suregry

CONTACTS AND LOCATIONS:
Overall Officials: ali ben ali, PROFESSOR, Study Director — university of sousse

IPD SHARING:
Plan to Share IPD: Undecided